CLINICAL TRIAL: NCT03718741
Title: Prospective Study of Adjuvant Radiotherapy in High Risk Bladder Cancer.
Acronym: Bladder-Aid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: few patients enrolled
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Head of Clinical Trials Department, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2107
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Adiuvant Radiotherapy +/- CT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adiuvant Radiotherapy +/- CT (Experimental): The radiation treatment will be delivered with two possible schedules, according to the presence of positive margins on the pathology specimen:
  * R0: PTVb + PTVn 50 Gy in 25 fractions
  * R1-2: PTVn 50 Gy in 25 fractions. PTVb (including cystectomy bed and residual tumor when present) 55 Gy in 25 fractions with simultaneous integrated boost (SIB).
  Considering an alfa/beta of 10 for bladder tumor and 3 for healthy tissues the equivalent doses will be respectively:
  BED10: 60/67.1; EQD2: 50/55.92 Gy BED3: 83.33/95.33; EQD2: 50/57.20 Gy
  Patients with ECOG PS<2, good haematological, hepatic and renal function (haemoglobin, neutrophil count, platelets, creatinine, glycaemia, Bilirubin, AST, ALT values within the limits of normal), will be submitted to concurrent cisplatin based weekly chemotherapy, 20-30 mg/m2, if they have not received neoadjuvant chemotherapy before surgery.
  Interventions: Radiation: Radiotherapy +/- CT

INTERVENTIONS:
Radiation: Radiotherapy +/- CT — Adiuvant Radiotherapy +/- weekly cisplatin

SUMMARY:
This prospective interventional study aims at evaluating the safety and efficacy of an adjuvant radiation treatment in cases of muscle-invasive bladder cancer, submitted to radical cystectomy and presenting clinic-pathological characteristics of high risk of recurrence.

DETAILED DESCRIPTION:
Bladder cancer represents the ninth neoplasm in the world, with approximately 430,000 new cases diagnosed in 2012. Of them, around 118,000 were diagnosed in Europe, and 52,000 had died from this disease.

Patients with advanced bladder cancer (stage ≥pT3) have a five-year overall survival of ~50% after cystectomy and pelvic lymphadenectomy +/- chemotherapy with approximately half of recurrences in the pelvis, either as isolated failures or synchronous with distant metastases. In fact, radical cystectomy with or without chemotherapy has a 5-year overall survival of approximately 60% for patients with pathologic T2 disease confined to the bladder but only 10-40% for stage ≥pT3 when disease extends into the extravesicular tissues.

Pelvic failures after radical cystectomy are common, especially for ≥pT3 urothelial carcinoma with a cumulative incidence of locoregional failure of 32% at 5 years in the SWOG 8710 cohort. Adjuvant radiation therapy (RT) can reduce locoregional failure and may even improve overall survival, but currently has no defined role, in part because of toxicity reported in older series using 1980s radiation techniques.

An externally validated risk stratification to identify patients at highest risk for local-regional failure who are most likely to benefit from adjuvant RT has been developed based on pathologic T-stage, surgical margin status, and extent of the lymph node dissection.

Local-regional recurrence following radical cystectomy for patients with locally advanced urothelial carcinoma is common. The risk of local-regional recurrence is not diminished with chemotherapy, and salvage treatment is rarely successful. Adjuvant RT can reduce locoregional failure and may even improve overall survival, but currently has no defined role, in part because of toxicity reported in older series using 1980s radiation techniques. Several lines of evidence support the hypothesis that improved local control may lead to improved disease-free and overall survival.

This prospective interventional study aims at evaluating the safety and efficacy of an adjuvant radiation treatment in cases of muscle-invasive bladder cancer, submitted to radical cystectomy and presenting clinic-pathological characteristics of high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Karnofsky index > 60 % (ECOG < 2)
* Histologically confirmed muscle-invasive bladder cancer (MIBC) submitted to radical cystectomy.
* Pathological T-stage > pT3, and/or pathological N-stage > pN1, and/or residual tumor present after surgery (R>1)
* No distant metastases
* Written informed consent

Exclusion Criteria:

* Prior RT in the pelvic region
* Presence of distant metastases
* Pregnancy
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Local Control Rate | 2 year
  This prospective interventional study aims at evaluating the safety and efficacy of an adjuvant radiation treatment in cases of muscle-invasive bladder cancer, submitted to radical cystectomy and presenting clinic-pathological characteristics of high risk of recurrence.

SECONDARY OUTCOMES:
PFS | 2 years
  Progression Free Survival
OS | 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No